CLINICAL TRIAL: NCT02018510
Title: A Phase 1, Open Label, Dose-escalation Study of the Safety, Pharmacokinetics and Antiretroviral Activity of 3BNC117 Monoclonal Antibody in HIV-infected and HIV-uninfected Volunteers
Brief Title: A Phase 1, Open Label, Dose-escalation Study of the Safety, Pharmacokinetics and Antiretroviral Activity of 3BNC117
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rockefeller University (Other)
Collaborators: Weill Medical College of Cornell University (Other); Brigham and Women's Hospital (Other); University of Cologne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MCA-0835
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Last update posted 2016-12-26 (Estimated); Status verified 2016-12

CONDITIONS: Healthy; HIV
Keywords: Healthy Volunteers; HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (15):
- Group 1A (Experimental): HIV-uninfected individuals
  1 mg/kg, single dose IV administration of 3BNC117
  Interventions: Biological: 1 mg/kg, single dose IV administration of 3BNC117
- Groups 1B (Experimental): HIV-uninfected individuals 3 mg/kg, single dose IV administration of 3BNC117
  Interventions: Biological: 3 mg/kg, single dose IV administration of 3BNC117
- Group 1C (Experimental): HIV-uninfected individuals 10 mg/kg, single dose IV administration of 3BNC117
  Interventions: Biological: 10 mg/kg, single dose IV administration of 3BNC117
- Group 1D (Experimental): HIV-uninfected individuals 10 mg/kg, two doses IV of 3BNC117
  Interventions: Biological: 10 mg/kg, two doses IV of 3BNC117
- Group 1E (Experimental): HIV-uninfected individuals 30 mg/kg, single dose IV administration of 3BNC117
  Interventions: Biological: 30 mg/kg, single dose IV administration of 3BNC117
- Group 1F (Experimental): HIV-uninfected individuals 30 mg/kg, two doses IV of 3BNC117
  Interventions: Biological: 30 mg/kg, two doses IV of 3BNC117
- Group 2A (Experimental): HIV-infected individuals on or off ART
  1 mg/kg, single dose IV administration of 3BNC117
  Interventions: Biological: 1 mg/kg, single dose IV administration of 3BNC117
- Group 2B (Experimental): HIV-infected individuals on or off ART 3 mg/kg, single dose IV administration of 3BNC117
  Interventions: Biological: 3 mg/kg, single dose IV administration of 3BNC117
- Group 2C (Experimental): HIV-infected individuals on or off ART 10 mg/kg, single dose IV administration of 3BNC117
  Interventions: Biological: 10 mg/kg, single dose IV administration of 3BNC117
- Group 2D (Experimental): HIV-infected individuals on or off ART 30 mg/kg, single dose IV administration of 3BNC117
  Interventions: Biological: 30 mg/kg, single dose IV administration of 3BNC117
- Group 2E (Experimental): HIV-infected individuals off ART, VL 2,000-100,000 copies/ml 30 mg/kg, single dose IV administration of 3BNC117
  Interventions: Biological: 30 mg/kg, single dose IV administration of 3BNC117
- Group 3 (Experimental): HIV-infected individuals off ART, VL < 2,000 copies/ml 30 mg/kg, single dose IV administration of 3BNC117
  Interventions: Biological: 30 mg/kg, single dose IV administration of 3BNC117
- Group 4 (Experimental): HIV-infected individuals on ART, VL < 100,000 copies/ml 30 mg/kg, single dose IV administration of 3BNC117
  Interventions: Biological: 30 mg/kg, single dose IV administration of 3BNC117
- Group 5A (Experimental): HIV-infected individuals on ART, VL < 20 copies/ml 10 mg/kg, single dose IV administration of 3BNC117
  Interventions: Biological: 10 mg/kg, single dose IV administration of 3BNC117
- Group 5B (Experimental): HIV-infected individuals on ART, VL < 20 copies/ml 30 mg/kg, single dose IV administration of 3BNC117
  Interventions: Biological: 30 mg/kg, single dose IV administration of 3BNC117

INTERVENTIONS:
Biological: 1 mg/kg, single dose IV administration of 3BNC117 — 1 mg/kg, single dose IV administration of 3BNC117
  Arms: Group 1A; Group 2A
Biological: 3 mg/kg, single dose IV administration of 3BNC117 — 3 mg/kg, single dose IV administration of 3BNC117
  Arms: Group 2B; Groups 1B
Biological: 10 mg/kg, single dose IV administration of 3BNC117 — 10 mg/kg, single dose IV administration of 3BNC117
  Arms: Group 1C; Group 2C; Group 5A
Biological: 30 mg/kg, single dose IV administration of 3BNC117 — 30 mg/kg, single dose IV administration of 3BNC117
  Arms: Group 1E; Group 2D; Group 2E; Group 3; Group 4; Group 5B
Biological: 10 mg/kg, two doses IV of 3BNC117 — 10 mg/kg, two IV administrations of 3BNC117 at weeks 0 and 12
  Arms: Group 1D
Biological: 30 mg/kg, two doses IV of 3BNC117 — 30 mg/kg, two IV administrations of 3BNC117 at weeks 0 and 12
  Arms: Group 1F

SUMMARY:
The proposed study is a first-in-man phase I study that aims to evaluate the safety, tolerability and pharmacokinetics of 3BNC117 in HIV-infected and HIV-uninfected subjects, and its antiretroviral activity in HIV-infected subjects.

DETAILED DESCRIPTION:
In preclinical studies carried out in humanized mice and non-human primates, 3BNC117 alone or in combination with other neutralizing antibodies led to protection from HIV-1 or SHIV infection and also to sustained suppression of HIV-1 plasma viremia. The aims of this protocol are to evaluate the safety, tolerability and pharmacokinetics profile of 3BNC117 in both HIV-infected and HIV-uninfected subjects,and its antiretroviral activity in HIV-infected subjects.

ELIGIBILITY:
Inclusion Criteria:

* Group 1 (HIV-uninfected):

  * Adult males and females, age 18 to 65
  * Amenable to HIV risk reduction counseling and agrees to maintaining behavior consistent with low risk of HIV exposure;
  * If a sexually active male or female, participating in sexual activity that could lead to pregnancy, agrees to use an effective method of contraception throughout the study.
* Groups 2-5 (HIV-infected):

  * Age 18 to 65
  * HIV infection confirmed by ELISA and immunoblot
  * Groups 2A-D - on ART with HIV-1 plasma RNA levels below 100,000 copies/ml, or off ART for at least 8 weeks with HIV-1 plasma RNA level between 2,000-100,000 copies/ml by standard assays on 2 occasions at least 1 week apart;
  * Group 2E - Untreated HIV-infected (not on ART for at least 8 weeks): HIV-1 RNA plasma levels between 2,000 - 100,000 copies/ml;
  * Group 3 - Untreated HIV controllers (not on ART for at least 8 weeks): HIV-1 RNA plasma level of < 2,000 copies/ml by standard assays, on 2 occasions, at least 1 week apart, and ART-naive.
  * Group 4 - ART treated with HIV-1 RNA plasma level of > 20 copies/ml by standard assays on 2 occasions, at least 1 week apart, while on combination antiretroviral therapy;
  * Groups 5A and 5B - ART treated with HIV-1 RNA plasma level of < 20 copies/ml by standard assays on 2 occasions, at least 1 week apart, while on combination antiretroviral therapy;
  * Current CD4 cell count > 300 cells/µl
  * If sexually active male and female, participating in sexual activity that could lead to pregnancy, agrees to use an effective method of contraception throughout the study.

Exclusion criteria:

* Group 1 (HIV-uninfected):

  * Confirmed HIV-1 or HIV-2 infection;
  * History of immunodeficiency or autoimmune disease; use of systemic corticosteroids, immunosuppressive anti-cancer, or other medications considered significant by the trial physician within the last 6 months;
  * Any clinically significant acute or chronic medical condition that in the opinion of the investigator would preclude participation;
  * Within the 12 months prior to enrollment, the volunteer has a history of sexually transmitted disease;
  * Hepatitis B (surface antigen, HbsAg) or hepatitis C (HCV antibodies);
  * Laboratory abnormalities in the parameters listed below:

    * Absolute neutrophil count ≤ 2,000
    * Hemoglobin ≤ 12 gm/dL if female; ≤ 13.5 gm/dL if male
    * Platelet count ≤ 140,000
    * ALT ≥ 1.25 x ULN
    * AST ≥ 1.25 x ULN
    * Total bilirubin ≥ 1.1 ULN
    * Creatinine ≥ 1.1 x ULN
    * Coagulation parameters (PT, PTT, INR) ≥ 1.1 x ULN
  * Pregnancy or breastfeeding;
  * Any vaccination within 14 days prior to 3BNC117 administration;
  * Receipt of any experimental HIV vaccine in the past or monoclonal antibody therapy of any kind in the past;
  * Participation in another clinical study of an investigational product currently or within past 12 weeks, or expected participation during this study.
* Groups 2-5 (HIV-infected):

  * History of AIDS-defining illness
  * History of systemic corticosteroids, immunosuppressive anti-cancer, or other medications considered significant by the trial physician within the last 6 months;
  * Any clinically significant acute or chronic medical condition, other than HIV infection, that in the opinion of the investigator would preclude participation;
  * Hepatitis B (surface antigen, HbsAg) or hepatitis C (HCV antibodies);
  * Laboratory abnormalities in the parameters listed below:

    * Absolute neutrophil count ≤ 1,300
    * Hemoglobin ≤ 10 gm/dL
    * Platelet count ≤ 125,000
    * ALT ≥ 2.0 x ULN
    * AST ≥ 2.0 x ULN
    * Total bilirubin ≥ 1.1 ULN
    * Creatinine ≥ 1.1 x ULN
    * Coagulation parameters ≥ 1.1 x ULN;
  * Current antiretroviral regimen includes either maraviroc or enfuvirtide;
  * Pregnancy or breastfeeding;
  * Any vaccination within 14 days prior to 3BNC117 administration;
  * Receipt of any experimental HIV vaccine or monoclonal antibody therapy of any kind in the past;
  * Participation in another clinical study of an investigational product currently or within past 12 weeks, or expected participation during this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 24 weeks
  To evaluate the safety and tolerability profile of one or two intravenous infusions of 3BNC117 at 3 increasing dose levels in HIV-infected and HIV-uninfected individuals.

SECONDARY OUTCOMES:
Pharmacokinetic profile | 24 hours post infusion
  To determine the pharmacokinetic profile of one or two intravenous infusions of 3BNC117 in HIV-uninfected and HIV-infected subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Caskey, MD, Principal Investigator — Rockefeller Univesrity
Locations (4):
- United States (3):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - The Rockefeller University, New York, New York
  - Weill Cornell Medical Center, New York, New York
- University of Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schoofs T, Klein F, Braunschweig M, Kreider EF, Feldmann A, Nogueira L, Oliveira T, Lorenzi JC, Parrish EH, Learn GH, West AP Jr, Bjorkman PJ, Schlesinger SJ, Seaman MS, Czartoski J, McElrath MJ, Pfeifer N, Hahn BH, Caskey M, Nussenzweig MC. HIV-1 therapy with monoclonal antibody 3BNC117 elicits host immune responses against HIV-1. Science. 2016 May 20;352(6288):997-1001. doi: 10.1126/science.aaf0972. Epub 2016 May 5. PMID 27199429